CLINICAL TRIAL: NCT02427997
Title: Virtual Reality-treadmill Combined Intervention for Enhancing Mobility and Cognitive Function in Patients With Multiple Sclerosis
Brief Title: VR-treadmill Combined Intervention for Enhancing Mobility and Cognitive Function in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TASMC-15-NG-063-CTIL
Record Dates: First submitted 2015-03-15; First posted 2015-04-28 (Estimated); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Multiple Sclerosis
Keywords: Virtual Reality; Treadmill; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treadmill training with virtual reality (Experimental): The TT+VR patients (i.e., the experimental arm) will receive 18 sessions (3 times per week x 6 weeks) of training that will consist of walking on a treadmill while wearing a safety harness (without body weight support, recall Figure 1), and while being provided with feedback from the system.
  Interventions: Behavioral: Treadmill training with Virtual Reality
- Treadmill training alone (Active Comparator): TT alone will receive conventional treadmill training with no feedback from the system. They will train with a safety harness 18 sessions (3 times per week x 6 weeks).
  Interventions: Behavioral: Treadmill training

INTERVENTIONS:
Behavioral: Treadmill training with Virtual Reality — VR is defined in general as a "high-end-computer interface that involves real time simulation and interactions through multiple sensorial channels". The VR system to be used requires subjects to negotiate virtual obstacles while walking on a treadmill, in a safe environment. This dual task activity has large cognitive components such as information processing, planning, and attention while allowing for training in a more stimulating and enriching environment that includes both cognitive and motor components.
  Other Names: TT+VR
  Arms: Treadmill training with virtual reality
Behavioral: Treadmill training — The participants will walk on the treadmill, their gait speed over-ground will be measured at the beginning of each week of training. Progression will include increasing the duration of each of the walking bouts and increasing walking speed.
  Other Names: TT
  Arms: Treadmill training alone

SUMMARY:
A prospective, randomized controlled single-blind trial will test the hypotheses that a 6- week intervention that combines treadmill training (TT) with virtual reality (VR) significantly improves real-life, functional mobility and cognitive abilities, keys to health-related quality of life in patients with MS.

DETAILED DESCRIPTION:
A prospective, single blinded,randomized controlled trial with 6 month follow-up will be employed to investigate the effects of treadmill training augmented with virtual reality on patients with MS. The study will include 200 participants. Participants will be randomized to either the intervention or active comparator. The intervention group will receive 18 sessions of Treadmill Training with Virtual Reality (TT+VR) and the active control comparison will receive 18 training sessions of treadmill training alone (TT) without the VR simulation All interventions will be delivered by therapists trained in the standard protocols. All subjects will be trained 3 times a week for 6 weeks, each session will last approximately 45 minutes.Training progression will be based on increasing both motor and cognitive challenges, individualized to the participant's level of performance.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if:

* They are between 18-65 years of age.
* They have a confirmed diagnosis of relapsing remitting MS.
* They have a score between 2 and 6 on the Expanded Disability Status Scale (EDSS)
* They are free from dementia as determined using the Mini Mental State Exam (MMSE>=24)
* They can walk on the treadmill without partial body weight support harness for 5 minutes at their preferred walking speed; this is set as the smallest bout length at the start of training.
* They have no history of epileptic seizures.
* They have no MS exacerbation within the preceding 4 weeks, as determined by interview and medical notes review.
* They have stable MS disease treatments (e.g., last intake of steroids occurred at least 50 days before the enrolment, MS-specific drugs stable from at least 3 months, symptomatic drugs stable from at least 1 month before the enrolment).
* They have adequate hearing (as evaluated by the whisper test and adequate vision capabilities (as measured using a Snellen chart, 6.20 cut-off).
* They are willing to commit to treadmill training program week and participate in all of the assessments.
* They provide informed written consent and are willing to be randomized to any of the 2 study arms.

Exclusion Criteria:

* Patients will be excluded if:

  * They cannot follow safety or training instructions.
  * They have another neurological disorder, unstable cardiovascular disease, diabetes, lower limb arthritis, acute lower back or lower extremity pain, peripheral neuropathy, rheumatic or severe orthopaedic problems that may interfere with walking, or have diagnosed psychiatric problems.
  * They are pregnant.
  * They are undergoing any experimental drug or other kind of therapy.
  * Their medication regime is likely to change during the course of the study.
  * They are already participating in an intensive exercise program. The use of walking aids will not exclude participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Immediate change in gait speed | One week post intervention
  Gait speed will be assessed under usual and dual task conditions and while negotiating physical obstacles, using a sensorized 7 meter carpet (PKMAS) and wearable body fixed sensors. These measures will be compared to baseline performance
Number of correct answers in the oral version of the Symbol Digit Modalities Test | One week post intervention
  The SDMT measures sustained attention and cognitive processing speed, is responsive to change and intervention in MS, can be administered in a relatively short period of time (< 5 minutes), is largely resistant to practice effects, is valid and reliable in MS, and has been used in many clinical trials in MS. The SDMT involves matching numbers to corresponding symbols for 90 seconds and is a main component of the brief international cognitive assessment for MS (BICAMS). The number of correctly matched symbols is considered the outcome score. This test measures attention and visual spatial processing, and it is likely that the SDMT will change in response to the TT+VR, and not in response to TT. Indeed, SDMT has been associated with cognitive motor interference in patients with MS.

SECONDARY OUTCOMES:
The 25 feet walk test (25FWT) | One week post intervention
  The T25-FW is a quantitative mobility and leg function performance test based on a timed 25-walk. It is the first component of the MSFC to be administered at each visit. The patient is directed to one end of a clearly marked 25-foot course and is instructed to walk 25 feet as quickly as possible, but safely. The time is calculated from the initiation of the instruction to start and ends when the patient has reached the 25-foot mark. The task is immediately administered again by having the patient walk back the same distance. Patients may use assistive devices when doing this task.

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Karni, MD, Principal Investigator — TASMC
Locations (2):
- Motor Control Research Lab at the University of Illinois Urbana-Champaign, Urbana, Illinois, United States
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

REFERENCES:
- [Derived] Galperin I, Mirelman A, Schmitz-Hubsch T, Hsieh KL, Regev K, Karni A, Brozgol M, Cornejo Thumm P, Lynch SG, Paul F, Devos H, Sosnoff J, Hausdorff JM. Treadmill training with virtual reality to enhance gait and cognitive function among people with multiple sclerosis: a randomized controlled trial. J Neurol. 2023 Mar;270(3):1388-1401. doi: 10.1007/s00415-022-11469-1. Epub 2022 Nov 11. PMID 36357586